CLINICAL TRIAL: NCT04887441
Title: Allergology: Information, Data and Knowledge Organization
Acronym: ALLERGIDOC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: LERASS-CERIC Université Paul Valéry Montpellier 3 Motpellier (Unknown); Occitanie Region (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0253
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Food Allergy; Peanut Allergy
Keywords: Food allergy; peanuts; Oral Immunotherapy; efficacy; safety
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Digital technology is essential in the field of health, via connected objects, the medical Internet or even telemedicine; and the info-communication practices (ways of getting information and communicating) of the actors go through digital devices. In addition, at present, the mass of activity documents to be managed in healthcare establishments and an abundant supply of documentary resources in health, available on the Internet, lead to infobesity, information pollution, and work overload. These phenomena lead to an increase in the time spent searching for relevant information and even to the burnout of healthcare professionals. A contextualization of the information communication systems through which the practices of health professionals pass therefore seems necessary so that the tools for managing, extracting and organizing knowledge can support these actors in their work.

In the field of allergies, there are many players, and the information that is useful to them is abundant and heterogeneous. This study is based on the hypothesis that a knowledge organization model, developed from existing practices, could make it possible to obtain satisfactory results when searching for information, and be integrated into the daily practices of actors by linking up with other already existing systems and tools.

ELIGIBILITY:
Inclusion criteria:

* Professionals from the Allergy Unit (doctors, interns, paramedics, study coordinators), in total around 20-30 people.
* Observations will be conducted during their team meetings and will not impact their workflow.
* Subjects publishing information on allergy on public web sites

Exclusion criteria:

* Professional not willing to participate to the research.
* Users publishing information on private web sites or forums.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professional of the Allergy Unit of the University Hospital of Montpellier (France)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the ontology model | 24 months
  measure (a) the efficiency of the model developed in the target technology (technology-focused evaluation), (b) the satisfaction of the professionals of the unit (user-focused evaluation) and (c) we will evaluate its formalization by an expert in knowledge organization systems (ontology-focused evaluation). The evaluations (a) and (b) will be made through the integration of the model into a future information communication device, and probably, into another existing device. The task will consist, for example, in the search for information and documents necessary for the information activities of professionals.

SECONDARY OUTCOMES:
Assessment and validation of the model | 18 months
  (a) At the end of the interrogation of a tool designed by professionals, we will calculate the recall rate, precision and F-measure. The efficiency of the model will be considered satisfactory, if the result obtained is equal or superior to other projects (b) The organizational model assessment will engage 10 professionals from the allergology unit. Professionals will assign (anonymously) the marks according to the level of satisfaction of the results of their request: 5 - Very satisfactory, 4 - Satisfactory, 3 - Fairly satisfactory, 2 - Unsatisfactory, 1 - Unsatisfactory. (c) The model will also be evaluated by a knowledge organization systems expert, selected from members of the International Society for Knowledge Organization.

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC